CLINICAL TRIAL: NCT02267213
Title: An Open-Label, Single-Arm, Two-Stage, Multi-Centre Phase II Study to Evaluate the Efficacy and Safety of TLC388 as Second-line Treatment in Subjects With Advanced Hepatocellular Carcinoma
Brief Title: Efficacy and Safety Study of TLC388 to Advanced Hepatocellular Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Current study design couldn't support futher development on this indication
Sponsor: Taiwan Liposome Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TLC388.4
Record Dates: First submitted 2014-09-11; First posted 2014-10-17 (Estimated); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — TLC 388

ARMS (1):
- Lipotecan (Experimental): Administer 40mg of Lipotecan at D1, D8, D15 of each cycles.
  Interventions: Drug: Lipotecan

INTERVENTIONS:
Drug: Lipotecan — Administer 40mg Lipotecan at D1, D8, D15 of each cycle.
  Other Names: Lipotecan, TLC388

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of TLC388 (Lipotecan) as a second line treatment in subjects with advanced Hepatocellular Carcinoma.

DETAILED DESCRIPTION:
A Phase II, open-label, single-arm, two-stage, multicenter study to evaluate the efficacy and safety of Lipotecan® monotherapy in patients with advanced hepatocellular carcinoma (HCC) and had failed sorafenib treatment due to sorafenib intolerance or radiographic progressive disease (PD).

Eligible patients received 40 mg/m2 of Lipotecan®, given as a 30-minute (+3 minutes) intravenous infusion, on Days 1, 8, and 15 of a 28-day cycle for maximum 6 cycles. Inter-cycle and intra-cycle dose delays were allowed within 21 days of the scheduled date to be reduced to 35 mg/m2 and further to 30 mg/m2 if a treatment-related adverse event (TRAE) met the criteria for dose reduction.

Tumor response was assessed every 2 cycles until Cycle 6, or at the early termination according to RECIST Version 1.1 judged by site investigator. The favorable response of CR, PR or SD would be confirmed within 28-35 days. Safety evaluations were conducted on a weekly basis from the day study treatment administered throughout each cycle.

ELIGIBILITY:
Inclusion Criteria:

* Radiological diagnosis of hepatic tumor(s) by contrast-enhanced study
* Subjects with advanced HCC who are not eligible for surgical resection or loco-regional therapy.
* Subjects with sorafenib treatment failure due to sorafenib intolerance or radiographic PD (as per RECIST v1.1). Prior sorafenib use should be ≥ 400 mg/day for at least 14 days.
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 1
* Child Pugh Score ≤ 6;
* A life expectancy of at least 12 weeks or more

Exclusion Criteria:

* Subjects who have received any systemic target therapy or systemic chemotherapy other than sorafenib for the treatment of HCC.
* Subjects who have received sorafenib within 2 weeks prior to the initiation of the treatment dose, or have any sorafenib-related toxicities not yet resolved to grade 1 or baseline.
* Subjects who have undergone liver transplantation surgery.
* Major surgery within 4 weeks prior to the initiation of the treatment dose (excluding implantation of the intravenous infusion device). Percutaneous liver puncture within 2 weeks prior to the initiation of the treatment dose.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2014-04-10 (Actual); Primary Completion 2015-07-09 (Actual); Study Completion 2015-07-09 (Actual)

PRIMARY OUTCOMES:
Disease Control Rate (DCR) | 8 weeks from initial treatment
  DCR (Disease control rate), the percentage of subjects with a best response rate of complete response (CR), partial response (PR), or stable disease (SD)

SECONDARY OUTCOMES:
Objective response rate (ORR; where ORR= CR rate + PR rate) | 8 weeks(Cycle 2), 16 weeks (Cycle 4), 24 weeks (Cycle 6) from initial treatment and/or Early termination (before 24 weeks)
  ORR (Objective response rate)
Duration of Disease control (DDC) | 2 months (Cycle 2), 4 months (Cycle 4) and 6 months (Cycle 6) and/or Early termination (before 6 months)
  Duration of disease control is defined as the time from first documented evidence of CR or PR or SD until the first documentation of PD or death due to any cause, whichever occurs first.
Time to Progression (TTP) | 2 months (Cycle 2), 4 months (Cycle 4) and 6 months (Cycle 6) and/or Early termination (before 6 months)
  Time to tumor progression is defined as the time from first study drug administration until the first documentation of tumor progression.
Progression Free Survival (PFS) | 2 months (Cycle 2), 4 months (Cycle 4) and 6 months (Cycle 6) and/or Early termination (before 6 months)
  The PFS is defined as the time from the first dose to the date of progression or death, whichever occurs first, and subjects with no evidence of progression or death at the time of study completion (the analysis cut-off date) or who are receiving any further anticancer therapy will be censored on the date of the last adequate tumor assessment.
Overall Survival (OS) | Up to 2 years from the last treatment of the last subject
  The OS is defined as the time from the first dose to the date of death, regardless of the cause of death, and subjects who are alive at the time of study completion will be censored at the last known alive date. Subjects who commence treatment with another anticancer agent will be censored at the day before the other anticancer treatment starts.
Change of Tumor markers/Bio-markers | Baseline, the first dose (Cycle 1 Day 1), 2 months(C2D1), 3 months(C3D1), 4 months(C4D1), 5 months(C5D1), 6 months(C6D1) and/or Early termination (before 6 months)
  tumor markers/biomarkers, including α-fetoprotein (AFP), vascular endothelial growth factor (VEGF), transforming growth factor-β1 (TGF-β1), and interleukin-6 (IL-6)
AEs | From ICF singed to 30 days after EOT
  Serious/ Adverse Events
Vital signs | Baseline, first treatment(C1D1), 1, 2, 4, 5, 6, 8, 9, 10, 12, 13, 14, 16, 17, 18, 20, 21, 22 weeks from the first treatment and/or Early termination (up to 24 weeks)
  evaluate at every administration and the end of treatment
Resting 12-lead ECGs | Baseline, the first dose (Cycle 1 Day 1), 2 months(C2D1), 3 months(C3D1), 4 months(C4D1), 5 months(C5D1), 6 months(C6D1) and/or Early termination (before 6 months)
  12-Lead ECGs
Hematology | Baseline, first treatment(C1D1), 1, 2, 4, 5, 6, 8, 9, 10, 12, 13, 14, 16, 17, 18, 20, 21, 22 weeks from the first treatment and/or Early termination (up to 24 weeks)
  evaluate at every administration and the end of treatment
Clinical chemistry | Baseline, first treatment(C1D1), 1, 2, 4, 5, 6, 8, 9, 10, 12, 13, 14, 16, 17, 18, 20, 21, 22 weeks from the first treatment and/or Early termination (up to 24 weeks)
  evaluate at every administration and the end of treatment
Urinalysis data | The first dose (Cycle 1 Day 1), 2 months(C2D1), 3 months(C3D1), 4 months(C4D1), 5 months(C5D1), 6 months(C6D1) and/or Early termination (before 6 months)
  Urinalysis Lab Values
PK parameters, including AUC, Cmax and Tmax of S,S-TLC388, S,R-TLC388, metabolites TLC-U1, TLC-U2, and topotecan | 0, 15, 29, 33, 40, 50 minutes, and 1, 1.5, 2, 4, 8 hour after the start of infusion of the 1st treatment and 1 week (2nd treatment); 0, 29 minutes and 4 hour after the start of infusion of the 3, 5, 6 and 7 weeks (the 3rd, 4th, 5th, 6th treatment)
  PK parameters

CONTACTS AND LOCATIONS:
Overall Officials: Yunlong Tseng, Study Director — Taiwan Liposome Company
Locations (12):
- China (4):
  - 307 Hospital of PLA, Beijin
  - Nanjing Bayi Hospital, Nanjing
  - Shanghai Cancer Hospital, Fudan University, Shanghai
  - Zhongshan Hospital, Fudan University, Shanghai
- Taiwan (8):
  - Chiayi Chang Gung Memorial Hosipital, Chiayi City
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - China Medical University Hosipital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Mackay Memorial Hosipital, Taipei
  - National Taiwan University Hosipital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - LinKou Chang Gung Memorial Hosipital, Taoyuan District